CLINICAL TRIAL: NCT05873465
Title: Effects of Cannabis Use on Sedation Requirements for Oral Surgery Procedures
Brief Title: Cannabis Use on Sedation for Oral Surgery Procedures
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15416
Record Dates: First submitted 2023-03-13; First posted 2023-05-24 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Cannabis Use
MeSH Terms: interventions — Midazolam; Fentanyl; Propofol; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Non-users (Active Comparator): Patients that don't use cannabis and will be submitted to sedation.
  Interventions: Drug: Sedation with Midazolam, Fentanyl, and Propofol; Procedure: Extraction of teeth
- Users that will stop use 72h before the procedure (Experimental): Patients that use cannabis and will stop using 72 hours before sedation.
  Interventions: Drug: Sedation with Midazolam, Fentanyl, and Propofol; Procedure: Extraction of teeth
- Users that will stop use 12h before the procedure (Experimental): Patients that use cannabis and will stop using 12 hours before sedation.
  Interventions: Drug: Sedation with Midazolam, Fentanyl, and Propofol; Procedure: Extraction of teeth

INTERVENTIONS:
Drug: Sedation with Midazolam, Fentanyl, and Propofol — Patients will have teeth extracted under sedation with Midazolam, Fentanyl, and Propofol
  Other Names: Sedation
Procedure: Extraction of teeth — The necessary teeth will be extracted
  Other Names: Surgical procedure

SUMMARY:
The use of Cannabis is increasing in the population, and the effects that this might have on different medical procedures are poorly understood. Particularly when submitted to deep sedation or general anesthesia, there is no consensus on best drugs or doses to deliver. The purpose of this clinical trial is to clarify the influence of chronic cannabis use during office based general anesthesia for extraction of teeth. The procedures will be performed in the Oral and Maxillofacial Surgery Clinic at the College of Dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years of age
* Class I or II according to the American Society of Anesthesiology (ASA)
* Need for dental extractions
* Extraction procedures with similar level of complexity

Exclusion Criteria:

* Surgical time lesser than 10 or greater than 30 minutes
* ASA status of III or greater
* BMI greater than 30 k/m2
* Pregnancy
* Use of anti-depressants, sedatives, or other mood-altering medications
* History of illicit substance abuse, alcoholism, or chronic opioid use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Propofol dose in milligrams | During the procedure
  Compare the total amount of propofol necessary to sedate patients that use cannabis with patients that do not use

SECONDARY OUTCOMES:
Heart rate in beats per minute | During the procedure
  Compare how the heart rate behave during the procedure in each group
Blood pressure in millimeters of mercury | During the procedure
  Compare how the blood pressure behave during the procedure in each group
Quality of sedation grading from 0 to 6 according to the Observer's Assessment of Alertness/Sedation scale | During the procedure
  Compare the difference in sedation quality during the procedure in each group

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, Oklahoma City, Oklahoma, United States